CLINICAL TRIAL: NCT00671723
Title: Dornase Alpha Versus Hypertonic Saline for Lung Atelectasis
Brief Title: Dornase Alpha Versus Hypertonic Saline for Lung Atelectasis in Non-Cystic Fibrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12783
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Atelectasis
Keywords: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Saline Solution; Saline Solution, Hypertonic; dornase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal saline (Placebo Comparator): Nebulized isotonic saline solution (4 ml of 0.9 % NaCl) twice daily, for a fixed period of 15 min, after a 15 min premedication with nebulized albuterol (2.5 mg diluted in 3 ml of 0.9 % NaCl).
  Interventions: Drug: Normal saline:
- Hypertonic saline (Active Comparator): Nebulized hypertonic saline solution (4 ml of 7 % NaCl) twice daily, for a fixed period of 15 min, after a 15 min premedication with nebulized albuterol (2.5 mg diluted in 3 ml of 0.9 % NaCl).
  Interventions: Drug: Hypertonic Saline
- Dornase alpha (Active Comparator): 2.5 mg of DNase (Dornase alpha, PULMOZYME® , Genentech, South San Francisco, CA), nebulized twice daily, after a 15 min premedication with nebulized albuterol (2.5 mg diluted in 3 ml of 0.9 % NaCl).
  Interventions: Drug: Dornase alpha

INTERVENTIONS:
Drug: Normal saline: — Nebulized isotonic saline solution (4 ml of 0.9 % NaCl) twice daily, for a fixed period of 15 min, after a 15 min premedication with nebulized albuterol (2.5 mg diluted in 3 ml of 0.9 % NaCl).
  Other Names: Normal Saline
  Arms: Normal saline
Drug: Hypertonic Saline — Nebulized hypertonic saline solution (4 ml of 7 % NaCl) twice daily, for a fixed period of 15 min, after a 15 min premedication with nebulized albuterol (2.5 mg diluted in 3 ml of 0.9 % NaCl).
  Arms: Hypertonic saline
Drug: Dornase alpha — 2.5 mg of DNase (Dornase alpha, PULMOZYME® , Genentech, South San Francisco, CA), nebulized twice daily, after a 15 min premedication with nebulized albuterol (2.5 mg diluted in 3 ml of 0.9 % NaCl).
  Arms: Dornase alpha

SUMMARY:
Despite the lack of trials proving the efficacy of DNase in non cystic fibrosis patients, it is currently heavily used in this population. In fact, per evidence of barcode scanning via Meditech computer system at OU Medical Center 93% of the DNase prescribed in 2005 was for non Cystic fibrosis patients with an estimated yearly cost of $341,968.15.In vitro studies showed that the effect of Dnase was minimal on sputum viscosity when compared to Hypertonic saline . Furthermore recent studies on hypertonic saline in cystic fibrosis patients showed that it is an inexpensive and safe therapy when preceded by a bronchodilator in patients with cystic fibrosis.

We hereby propose a prospective randomized trial to compare the efficacy of hypertonic saline, DNase, vs. normal saline in the treatment of atelectasis in non cystic fibrosis, mechanically ventilated patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patient on invasive mechanical ventilation
2. New Onset (<48 hours) lobar or multilobar lung atelectasis based on CXR

Exclusion Criteria:

1. Asthma
2. Severe COPD (FEV1<30%)
3. Pneumothorax or massive pleural effusion, thought to be causing the atelectasis
4. Lobar atelectasis secondary to compressive tumor.
5. Severe hypoxemia (PaO2/FiO2 < 75)
6. Hemodynamic Instability
7. Cystic fibrosis patients
8. Allergy to DNase
9. Patients on Acetylcysteine
10. Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Keddissi, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Presbyterian Hospital, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Youness HA, Mathews K, Elya MK, Kinasewitz GT, Keddissi JI. Dornase alpha compared to hypertonic saline for lung atelectasis in critically ill patients. J Aerosol Med Pulm Drug Deliv. 2012 Dec;25(6):342-8. doi: 10.1089/jamp.2011.0954. Epub 2012 Mar 13. PMID 22413805

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Saline | Hypertonic Saline | Dornase Alpha
Started | 11 | 11 | 11
Completed | 11 | 11 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Mechanically ventilated patients with new onset ( < 48 h) lobar or multilobar atelectasis
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Hypertonic Saline | Dornase Alpha | Total
Number analyzed (Participants) | 11 | 11 | 11 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (15) | 48 (15) | 49 (18) | 47 (16)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 9 | 29
  >=65 years | 2 | 0 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 8 | 7 | 7 | 22
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in the Chest X-ray Atelectasis Score
Description: Each CXR was assigned an atelectasis score.(*) The absence or presence of contralateral hyperinflation was marked as 0 or 1 point, respectively. The absence or presence of mediastinal shift was scored as 0 or 1, respectively. Atelectasis was scored for each lobe. A partial atelectasis of one lobe was scored as one point, whereas complete atelectasis of a lobe was marked as two points. The distinction between infiltrate and atelectasis as well as the total scoring was done by the interpreting radiologist. These results were summed for each CXR. The score range from 0 to 10 with 0 indicates "no atelectasis",higher value indicates progressively more atelectasis.
  *Hendriks T, de Hoog M, Lequin MH, Devos AS, and Merkus PJ: DNase and atelectasis in non-cystic fibrosis pediatric patients. Crit Care. 2005;9:R351-R356.
Time Frame: Baseline(Day 0) to Day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | Hypertonic Saline | Dornase Alpha
Number analyzed (Participants) | 11 | 11 | 11
units on a scale | -1 (2.12) | -0.86 (1.34) | -2.18 (1.33)

2. Secondary Outcome: Rate of Extubation
Description: percentage of patient who were extubated at day 7
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | Hypertonic Saline | Dornase Alpha
Number analyzed (Participants) | 11 | 11 | 11
Participants | 6 | 5 | 7

ADVERSE EVENTS:
Arm/Group | Normal Saline | Hypertonic Saline | Dornase Alpha
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes